CLINICAL TRIAL: NCT02016547
Title: Thrombectomy Under Reopro Versus Alteplase and Neurologic Deficit Outcome Trial
Brief Title: Thrombectomy Under Reopro Versus Alteplase to Treat Stoke
Acronym: TURANDOT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: SOS Attaque Cérébrale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-005493-66
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Infarction, Middle Cerebral Artery
Keywords: Stroke; Middle Cerebral Artery; Thrombectomy; Mechanical Thrombolysis; Abciximab
MeSH Terms: conditions — Infarction, Middle Cerebral Artery; Stroke | interventions — Thrombectomy; Tissue Plasminogen Activator; Infusions, Intravenous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- abciximab IV and thrombectomy (Experimental): abciximab IV (0.25mg/kg by IV bolus, following by 0.125μg/kg by 12 hours IV drip) and thrombectomy
  Interventions: Procedure: abciximab IV and thrombectomy
- alteplase (Active Comparator): alteplase 0.9mg/kg (10% by IV bolus following by 90% by 1 hour IV drip)
  Interventions: Drug: alteplase 0.9mg/kg (10% by IV bolus following by 90% by 1 hour IV drip)

INTERVENTIONS:
Procedure: abciximab IV and thrombectomy
  Arms: abciximab IV and thrombectomy
Drug: alteplase 0.9mg/kg (10% by IV bolus following by 90% by 1 hour IV drip)
  Arms: alteplase

SUMMARY:
Intravenous (IV) Alteplase (rt-PA) is the gold standard for brain infarction within 4 h 30 of symptoms onset. Efficacy of this therapy is limited in the setting of large artery occlusions. For middle cerebral artery occlusions (MCA)or internal carotid artery occlusions (ICA), recanalization rates will drop as low as 10%. This element is critical as prognosis is linked to recanalization. Arterial re-occlusions are frequent and may reach 30%, which limits IV thrombolysis efficacy.With the endovascular approach, recanalization rates may reach 90% with last generation devices. A recent meta-analysis has shown that the best candidates for thrombectomy are MCA occlusions. In the coronary literature, endovascular therapy efficacy is increased in association with antiplatelets such as abciximab. The aim of the study was to assess the feasibility of thrombectomy associated with abciximab on revascularisation (TICI score), as well as safety (symptomatic intracranial bleeding), in order to design a clinical trial versus the gold standard for acute ischemic stroke revascularization strategies using IV rt-PA.This is a controlled, pilot study, evaluating feasibility and safety of thrombectomy with abciximab versus IV rt-PA in acute ischemic stroke patients within 4h30 of symptoms onset.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs consistent with acute ischemic stroke < 4.5 hours
* Cerebral infarction and middle cerebral artery occlusion, without any hemorrhage documented by MRI or CT
* 4 < National Institute of Health Stroke Score (NIHSS) < 25
* age > 18 years
* no prestroke functional dependance : modified Rankin score ≤ 2
* subject or subject's legally authorized representative has signed and dated an Informed Consent Form according to french regulations and ethic committee.

Exclusion Criteria:

* pregnant or lactating female
* coma (vigilance NIHSS > 1)
* epilepsy
* recent history of stroke
* anticoagulant therapy or International Normalized Ratio (INR) > 1.7 ; heparin therapy within past 24 hours and Temps de Cephaline Activee (TCA) extension
* previous subarachnoid hemorrhage or clinical presentation suggesting a subarachnoid hemorrhage, even if initial CT or MRI scan are normal
* known hereditary or acquired hemorrhagics diathesis, coagulation factor deficiency
* uncontrolled hypertension defined as systolic blood pressure ≥ 185 millimeters of mercury (mmHg) or diastolic blood pressure > 110 mmHg at time of admission and time of threat
* lumbar ar arterial puncture within past 7 days
* major surgery within past 2 months
* gastrointestinal hemorrhage or urinary hemorrhage
* myocardial infarction within past 21 days
* pericarditis within past 3 months
* suspicion of bacterial endocarditis within past 3 months
* previous of aortic dissection
* baseline lab values : TCA > 40, platelets < 100 000/mm3, glucose < 3 mmol/l or > 22 mmol/l
* hepatic insufficiency
* CT or MRI evidence oh hemorrhage
* CT or MRI evidence of mass effect or intra-cranial tumor
* CT showing hypodensity or MRI showing hyperdensity involving greater than 1/3 of the middle cerebral artery territory (ASPECT score < 7)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
recanalization rate | 24 hours

SECONDARY OUTCOMES:
Symptomatic intracranial bleeding | 24 hours
percentage of patients with a favorable outcome | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Stroke Center, Bichat Hospital, Paris, France